CLINICAL TRIAL: NCT05122702
Title: Efficacy and Safety of an Innovative Chinese Herbal Formula for the Treatment of Macular Edema: A Double-blind, Randomized, Placebo-Controlled Trial
Brief Title: An Innovative Chinese Herbal Formula for Macular Edema
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Prof. Lin Zhixiu, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Macular Edema study
Record Dates: First submitted 2021-07-23; First posted 2021-11-17 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Macula Edema

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Arm (Experimental): 18.75g of "Modified Shenling Baizhu San" granules will be taken twice daily for 12 weeks.
  Interventions: Drug: modified Shenling Baizhu San
- Placebo Arm (Placebo Comparator): 18.75g of placebo granules will be taken twice daily for 12 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: modified Shenling Baizhu San — modified Shenling Baizhu San granules, twice daily for 12 weeks.
  Arms: Active Arm
Other: Placebo — Placebo granules, twice daily for 12 weeks.
  Other Names: Placebo granules
  Arms: Placebo Arm

SUMMARY:
Macular edema (ME) is caused by hyperpermeability of retinal vessels and/or decreased efflux of fluid across the retinal pigment epithelium induced by outer/inner blood-retinal barrier dysfunction (BRB). It is most commonly seen following many diseases such as diabetes mellitus (DM), intraocular surgery, uveitis, retinal vein occlusion, and posterior segment inflammatory disease. An estimated 11% of patients with DM develop diabetic macular edema (DME). While the overall prevalence of DME among patients with DM aged 20 to 79 years is approximately 7.5%, the risk increases over time. Currently, there is no cure for ME.

Chinese medicine (CM) is widely used to manage ME in China and other East Asian countries. Among them, Shenling Baizhu San (SBS) is one of the most commonly used formulae. In this proposal, a randomized, double-blind, placebo-controlled, multicenter clinical trial will be undertaken to evaluate the efficacy and safety of modified SBS (mSBS) developed by the project team for the treatment of ME.

Eligible subjects will be recruited and assigned randomly to receive orally mSBS or placebo twice a day for 12 consecutive weeks, with follow-up for another 4 weeks after stopping the treatment to observe the duration of efficacy.

DETAILED DESCRIPTION:
Macular edema (ME) is characterized by hyperpermeability of retinal vessels and/or decreased efflux of fluid across the retinal pigment epithelium, and the condition can be induced by outer/inner blood-retinal barrier dysfunction (BRB). It is most commonly seen following a number of local and systemic diseases and procedures such as diabetes, intraocular surgery, uveitis, retinal vein occlusion, posterior segment inflammatory disease, and cataract surgery. Pathologically, ME is characterized by a retinal thickening in the macular area due to the breakdown of the BRB. ME patients often suffer from blurred vision, dark spots, and deformation, which can seriously affect their central vision, and in severe case, can lead to blindness.

Nowadays, ME treatment options include intravitreal anti-vascular endothelial growth factor (VEGF) agents, intravitreal long-acting steroid, non-steroidal anti-inflammatory drugs, corticosteroids, carbonic anhydrase inhibitors, and subthreshold macular laser. Although the above treatment options have made great progress, the possible side effects of the potentially toxic pharmaceutical agents should be always alert by clinician. A stepwise therapeutic approach is a challenge for the management of ME arises in the chronic and persistent case. Additionally, surgical management should be considered for unremitting cases of ME. Side effects such as scotomas, corresponding to the laser burns, have been frequently noticed by the patients following photocoagulation.

Currently, there is no cure for ME in conventional medicine. Chinese medicine (CM) is becoming popular for managing ME in China and other East Asian countries. Several research groups worldwide have previously conducted clinical studies to evaluate the effectiveness of Chinese herbal medicines for the treatment of ME in recent decades. This study is of an innovative Chinese herbal formula modified from a famous ancient formula for the treatment of macular edema. The goal of this treatment modality is to reduce the accumulation of intraretinal fluid, thus leading to improved visual acuity. Among different Chinese herbal formulae for ME, Shenling Baizhu San (SBS), which was originally described "Formulas from the Imperial Pharmacy" (Taiping Huiming Hejiju Fang in Chinese), has been reported have good efficacy in the treatment.

This study will use an innovative Chinese herbal formula modified from a famous ancient formula for the treatment of ME. This clinical study will be able to provide robust clinical evidence on the efficacy and safety of mSBS for ME. Subjects will be recruited and assigned to receive orally mSBS or placebo twice a day for 12 weeks, with follow-up for another 4 weeks after stopping the treatment to observe the duration of efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Both gender;
* Age from 18 to 80 years;
* Known diagnosed with ME;
* Agree to under optical examination and willing to complete questionnaires and take medications as scheduled; and
* Agree to participate in the study and provide written informed consent. (for those illiterate subjects, their family member can sign the consent form upon subject's agreement)

Exclusion Criteria:

* Known ocular media opacities, such as cataract, vitreous hemorrhage, asteroid hyalosis, that affect the determination of retinal thickness from OCT imaging;
* Known clinically significant macular edema (CSME). The definition of CSME: if one or more of the following criteria are met 1) retinal thickening at or within 500 μm of the center of the macula; 2) hard exudates at or within 500 μm of the center of the macula, if associated with adjacent retinal thickening; 3) a zone or zones of retinal thickening one disc area in size, at least part of which is within one disc diameter of the center of the macula;
* On concomitant oral or injectable corticosteroids, topical non-steroidal anti-inflammatory drugs (NSAID) eye drops, leukotriene inhibitors, anti-VEGF, immunosuppressants for the treatment of ME within past 6 months or other Chinese herbal medicine for the treatment of ME within past month;
* Impaired hematological profile and liver / renal function exceeds the upper limit of the reference value by 2 times;
* Documented pregnant or lactating; or
* Subjects participating in other clinical studies at the same time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-07-12 (Actual); Primary Completion 2024-07-31 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
The change of Central retinal (macular) thickness (CMT) score at week 12 | 12 weeks
  A standard nine-subfield Early Treatment of Diabetic Retinopathy Study grid will represent the averaged CMT and total macular volume. The highest score of CMT, the more severe of edema.
The change of Nest-Corrected Visual Acuity (BCVA) score at week 12 | 12 weeks
  For BCVA, Each letter of the acuity chart will score a value of 0.02 log unit. The highest score of central retinal (macular) thickness (CMT), the poorer of visual acuity.

SECONDARY OUTCOMES:
The change of Best-Corrected Visual Acuity (BCVA) score at week 16 | 16 weeks
  For BCVA, Each letter of the acuity chart will score a value of 0.02 log unit. The highest score of central retinal (macular) thickness (CMT), the poorer of visual acuity.
The change of Central retinal (macular) thickness (CMT) at week 16 | 16 weeks
  A standard nine-subfield Early Treatment of Diabetic Retinopathy Study grid will represent the averaged CMT and total macular volume. The highest score of CMT, the more severe of edema.
The change of Optical coherence tomography angiography (OCTA) at week 12 & 16 | 12 & 16 weeks
  OCTA will measured in both eyes of all participants. The highest score, the more severe of the angiography.
The change of Five-Level Version of EuroQoL-five dimensions questionnaire (EQ-5D-5L) at week 12 & 16 | 12 & 16 weeks
  It is a versatile quality of life (QOL) instrument with five dimensions used to calculate quality-adjusted life years.
The change of National Eye Institute Visual Functioning Questionnaire-25 (NEI-VFQ-25) at week 12 & 16 | 12 & 16 weeks
  It is a vision-specific measure of HRQoL composed of eight multi-item scales, four single-item scales, and one composite score ranging in value from 0 (poor) to 100 (high HRQoL).
Adverse event | 16 weeks
  Any adverse event related to study treatment will be analyzed throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Zhixiu Lin, PhD, Principal Investigator — Hong Kong Institute of Integrative Medicine
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No